CLINICAL TRIAL: NCT06811974
Title: Comparison of the Efficiency of Tissue Adhesive (Periacryl 90) and Silk Suture in Bilateral Mandibular Impacted Wisdom Dental Surgery
Brief Title: Comparison of the Efficiency of Tissue Adhesive (Periacryl 90) and Silk Suture in Mandibular Impacted Wisdom Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YYU-04/18.05.2022
Record Dates: First submitted 2025-01-24; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Impacted Mandibular Third Molar Extraction
Keywords: tissue adhesive; impacted wisdom tooth; silk suture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue adhesive (Periacryl 90) (Active Comparator): After the extraction of the impacted lower wisdom tooth, the wound area was closed using tissue adhesive.
  Interventions: Procedure: Impacted lower wisdom tooth extraction
- Silk suture (Active Comparator): After the extraction of the impacted lower wisdom tooth, the wound area was closed using silk sutures.
  Interventions: Procedure: Impacted lower wisdom tooth extraction

INTERVENTIONS:
Procedure: Impacted lower wisdom tooth extraction — One of the most frequently performed procedures in maxillofacial surgery is impacted wisdom tooth surgery. An impacted tooth is defined as a tooth that is not fully or partially erupted and is blocked from eruption by another tooth, bone, or soft tissue, and thus has a low probability of eruption. The tooth is blocked from eruption by adjacent hard or soft tissue, including bone or dense soft tissue. The most common complications after impacted wisdom tooth surgery are pain, edema, trismus, and alveolar osteitis.

SUMMARY:
In this study, bilateral It is aimed to compare the efficacy of tissue adhesive (Periacryl 90) and silk suture in mandibular impacted wisdom tooth surgery.

DETAILED DESCRIPTION:
In the study carried out on a total of 30 patients, 21 females and 9 males, 60 fully impacted lower wisdom teeth were extracted bilaterally and in the same position. One of the bilateral bilateral teeth of the patients was randomly selected and tissue adhesive (Periacryl 90) was applied for wound closure as the experimental group, while the other tooth was determined as the control group and the wound was closed with silk suture. The selected party was determined by the closed envelope method. After the first impacted tooth was extracted, it was waited until the wound healed and the symptoms disappeared completely, then the other tooth was extracted. In both tooth extractions, wound healing, edema and trismus were evaluated on the 3rd and 7th days. Wound healing was evaluated as good, acceptable and bad. VAS (Visual Analog Scale) was used for pain assessment and assessment was made at 3, 6, 12 and 24 hours and 2, 3, 4, 5, 6 and 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-35 years who accepted the study conditions and had bilateral, bone or mucosal retention, and completely impacted wisdom teeth in the similar position with an indication for extraction due to prophylactic or orthodontic treatment in the lower jaw were included in the study.

Exclusion Criteria:

* Individuals with any systemic disease
* Individuals with a history of allergy to the drugs to be used in the study
* Pregnant and breastfeeding individuals
* Individuals with pain, swelling or trismus in the last 10 days
* Individuals with different positions on the right and left sides
* Individuals who did not sign the voluntary consent form
* Individuals with pathology in the impacted tooth area
* Individuals with limited mouth opening

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Wound Healing | 3. and 7. days
  All patients were called for follow-up visits on the 3rd day and 1 week later and were examined by the same physician. During the follow-up visits, the status of wound healing was evaluated in 3 different statuses. These 3 statuses were recorded as good, acceptable and poor. Wound healing deteriorated from good to poor.
Edema | 3. and 7. days
  In order to evaluate edema, the distances between points marked extra orally in 5 different regions on the face were measured and recorded in mm (angulus-tragus point, angulus-lateral corner of the eye, angulus-nasal wing, angulus-lateral commissure, angulus-pogonion point).
Trismus | 3. and 7. days
  The evaluation of trismus was evaluated by measuring the mouth opening before the operation and also on the 3rd and 7th days after the operation. The patients were asked to open their mouths as much as possible and the distance between the incisal edges of the lower and upper central incisors was measured in millimeters with the help of a precision ruler. This process was repeated 3 times for each measurement and the arithmetic average of the values found was taken.
VAS Pain Scor | 3, 6, 12 and 24 hours and 2, 3, 4, 5, 6 and 7 days.
  VAS (Visual Analog Scale) was used for pain assessment. VAS pain assessment includes scores between 0 and 10. (0: no pain; 10: unbearable pain.) As the score increases, the pain worsens.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl Üniversitesi Diş Hekimliği Fakültesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bao Z, Gao M, Sun Y, Nian R, Xian M. The recent progress of tissue adhesives in design strategies, adhesive mechanism and applications. Mater Sci Eng C Mater Biol Appl. 2020 Jun;111:110796. doi: 10.1016/j.msec.2020.110796. Epub 2020 Mar 5. PMID 32279807
- [Background] Bamgbose BO, Akinwande JA, Adeyemo WL, Ladeinde AL, Arotiba GT, Ogunlewe MO. Effects of co-administered dexamethasone and diclofenac potassium on pain, swelling and trismus following third molar surgery. Head Face Med. 2005 Nov 7;1:11. doi: 10.1186/1746-160X-1-11. PMID 16274480
- [Background] Bal-Ozturk A, Cecen B, Avci-Adali M, Topkaya SN, Alarcin E, Yasayan G, Ethan YC, Bulkurcuoglu B, Akpek A, Avci H, Shi K, Shin SR, Hassan S. Tissue Adhesives: From Research to Clinical Translation. Nano Today. 2021 Feb;36:101049. doi: 10.1016/j.nantod.2020.101049. Epub 2020 Dec 20. PMID 33425002
- [Background] Ballestas SA, Turner TC, Kamalakar A, Stephenson YC, Willett NJ, Goudy SL, Botchwey EA. Improving hard palate wound healing using immune modulatory autotherapies. Acta Biomater. 2019 Jun;91:209-219. doi: 10.1016/j.actbio.2019.04.052. Epub 2019 Apr 25. PMID 31029828
- [Background] Asher R, Chacartchi T, Tandlich M, Shapira L, Polak D. Microbial accumulation on different suture materials following oral surgery: a randomized controlled study. Clin Oral Investig. 2019 Feb;23(2):559-565. doi: 10.1007/s00784-018-2476-0. Epub 2018 May 2. PMID 29717362
- [Background] Amiel GE, Sukhotnik I, Kawar B, Siplovich L. Use of N-butyl-2-cyanoacrylate in elective surgical incisions--longterm outcomes. J Am Coll Surg. 1999 Jul;189(1):21-5. doi: 10.1016/s1072-7515(99)00068-x. PMID 10401736
- [Background] American Academy of Pediatric Dentistry Ad Hoc Committee on Pedodontic Radiology; American Academy of Pediatric Dentistry Council on Clinical Affairs. Guideline on prescribing dental radiographs for infants, children, adolescents, and persons with special health care needs. Pediatr Dent. 2005-2006;27(7 Suppl):185-6. No abstract available. PMID 16541920
- [Background] Al-Moraissi EA, Al-Zendani EA, Al-Selwi AM. Efficacy of Submucosal Injection of Chymotrypsin, Oral Serratiopeptidase or Oral Dexamethasone in Reducing Postoperative Complications Following Impacted Lower Third Molar Surgery: A Prospective, Randomized, Double-Blind, Controlled Clinical Trial. Front Oral Health. 2020 Dec 8;1:575176. doi: 10.3389/froh.2020.575176. eCollection 2020. PMID 35047980
- [Background] Akbulut N, Ustuner E, Atakan C, Colok G. Comparison of the effect of naproxen, etodolac and diclofenac on postoperative sequels following third molar surgery: a randomised, double-blind, crossover study. Med Oral Patol Oral Cir Bucal. 2014 Mar 1;19(2):e149-56. doi: 10.4317/medoral.19518. PMID 24316711
- [Background] Ali AS, Benton JA, Yates JM. Risk of inferior alveolar nerve injury with coronectomy vs surgical extraction of mandibular third molars-A comparison of two techniques and review of the literature. J Oral Rehabil. 2018 Mar;45(3):250-257. doi: 10.1111/joor.12589. Epub 2017 Dec 11. PMID 29171914

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT06811974/Prot_SAP_000.pdf